CLINICAL TRIAL: NCT02046174
Title: A Phase IIb, Nonrandomized, Open-Label Trial With Mouse Renal Adenocarcinoma (RENCA) Cell Containing Agarose-Agarose Macrobeads Compared With Best Supportive Care in Patients With Treatment-Resistant, Metastatic Colorectal Carcinoma
Brief Title: Open-Label Phase IIb Efficacy Trial of Cancer Macrobeads Compared to Best Supportive Care in Colorectal Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Rogosin Institute (Other)
Collaborators: Vital Systems Inc. (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RI-MB-203; 1310014396 (Other: Weill Cornell Medical College IRB)
Record Dates: First submitted 2014-01-21; First posted 2014-01-27 (Estimated); Results first posted 2021-03-24 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-02

CONDITIONS: Colorectal Cancers
Keywords: colon; colorectal; rectal; cancer; macrobead; stage IV; metastatic; biological; mouse cells; new york; new jersey; clinical research
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Macrobead Implantation Arm (Experimental): patients who will undergo up to 4 implantations of RENCA macrobeads (no less than 3 months apart), at an amount of 8 RENCA macrobeads per kilogram of body weight
  Interventions: Biological: RENCA macrobeads
- Best Supportive Care Arm (No Intervention): patients who will receive, or continue receiving, best supportive care, defined as management of symptoms aimed at maintaining or improving quality of life, but not including approved therapies targeting the patient's malignancy

INTERVENTIONS:
Biological: RENCA macrobeads
  Other Names: mouse renal adenocarcinoma (RENCA) macrobeads; macrobead
  Arms: Macrobead Implantation Arm

SUMMARY:
This is a clinical research study of an investigational (FDA IND-BB 10091) treatment for patients with advanced colorectal cancer that no longer responds to standard therapies.

The treatment is being evaluated for its effect on tumor growth. It consists of the placement (implantation) of small beads that contain mouse renal adenocarcinoma cells (RENCA macrobeads). The cells in the macrobeads produce substances that have been shown to slow or stop the growth of tumors in experimental animals and veterinary patients. It has been tested in 31 human subjects with different types of cancers in a Phase I safety trial. Phase II studies in patients with colorectal, pancreatic or prostate cancers are in progress

DETAILED DESCRIPTION:
This is a Phase IIb, multicenter, nonrandomized, open-label study with RENCA macrobeads in patients with treatment-resistant, metastatic colorectal carcinoma to determine the effect of RENCA macrobead implantation on overall survival compared with best supportive care.

Two treatment groups will be enrolled in this study, as follows:

* Group A (n=40) - patients who will undergo up to 4 implantations of RENCA macrobeads (no less than 3 months apart), at a dosage level of 8 RENCA macrobeads per kilogram of body weight
* Group B (n=80) - patients who had previously decided (independently of this study) to receive, or continue receiving, best supportive care, defined as management of symptoms aimed at maintaining or improving quality of life, but not including approved therapies targeting the patient's malignancy

ELIGIBILITY:
Inclusion Criteria:

Patients in both treatment groups must meet all of the following criteria to be considered eligible to participate in the study:

* Adult men or women, aged 18 years or older, with histologically-confirmed, metastatic adenocarcinoma of the colon or rectum that has been proven to be resistant to available treatment options, including at least 2 such options from available chemotherapy, targeted, and/or other regimens.
* Radiographic evidence of disease progression.
* Life expectancy of at least 6 weeks, in the investigator's opinion, at the time disease progression is documented.
* Considered surgical candidates on the basis of co-morbidity risks, number and sites of metastases, and ability to undergo general anesthesia.
* Able to understand the risks of experimental therapy and provide written consent by signing the appropriate form.

Patients in Group A must also meet all of the following additional criteria:

* ECOG performance status score of 0, 1, or 2.
* Adequate hematologic function, defined as follows:

  1. absolute neutrophil count (ANC) ≥1500 /mL
  2. hemoglobin ≥9 g/dL
  3. platelets ≥75,000 /mL
* Adequate hepatic function, defined as follows:

  1. bilirubin ≤1.5 times the upper limit of normal (x ULN)
  2. aspartate transaminase (AST) ≤3 x ULN, or ≤5 x ULN if liver metastases are present
  3. alanine transaminase (ALT) ≤3, x ULN, or ≤5 x ULN if liver metastases are present
* Adequate renal function, defined as creatinine ≤2.0 mg/dL.
* Adequate coagulation function, defined as follows:

  1. International Normalized Ratio (INR) ≤1.5 or between 2 and 3 if the patient is receiving anticoagulation
  2. Partial Thromboplastin Time (PTT) ≤5 seconds above the ULN Note: Patients receiving full-dose anticoagulation therapy must have received a stable dose of oral anticoagulant therapy or low-molecular-weight heparin.
* Clinically significant toxic effects of chemotherapy (excluding alopecia), radiotherapy, hormonal therapy, or prior surgery must have resolved to Grade 1 or better, with the exception of peripheral neuropathy, which must have resolved to Grade 2 or better.
* Female participants of childbearing potential must have had a negative serum pregnancy test at screening; and must also agree to contraceptive use while on study if sexually active. Male subjects and their partners must have agreed to use condoms.

Exclusion Criteria:

Patients in either treatment group who meet any of the following criteria will be excluded from participating in the study:

* Hepatic blood flow abnormalities, i.e., portal vein hypertension and thrombosis, and/or a large volume of ascites.
* Concurrent cancer of any other type, except skin cancers other than melanoma.
* A positive test result for HIV or any hepatitis other than A at screening.
* Considered by the investigator to be unsuitable for participation in the study upon review of medical history, physical examination, or clinical laboratory test results.

Patients in Group A who meet any of the following criteria will be excluded from participating in the study:

* Received FDA-approved chemotherapy within 3 weeks of Day 0, or bevacizumab (or similar drugs) within 4 weeks of Day 0, or radiation therapy at any site within 4 weeks of Day 0.
* Investigational anticancer therapy within 4 weeks of Day 0.
* Positive reaction to the skin test for allergy to mouse antigen.
* History of hypersensitivity reaction that, in the opinion of the investigator, poses an increased risk of an allergic reaction to the RENCA macrobeads, particularly any known allergy to murine antigens or body tissues.
* Ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, serious cardiac arrhythmias (with the exception of well controlled atrial fibrillation), active bleeding, or psychiatric illness, or social situations that could interfere with the patient's ability to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2014-04-03 (Actual); Primary Completion 2018-10-22 (Actual); Study Completion 2018-10-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas J Fahey, III., M.D., Principal Investigator — Weill Cornell Medical Center / New York-Presbyterian Hospital
Locations (4):
- United States (4):
  - University of Kansas Cancer Center, Westwood, Kansas
  - Weill Cornell Medical Center / The Rogosin Institute, New York, New York
  - Calvary Hospital, The Bronx, New York
  - The Ohio State University; OSU Comprehensive Cancer Center, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Smith BH, Gazda LS, Conn BL, Jain K, Asina S, Levine DM, Parker TS, Laramore MA, Martis PC, Vinerean HV, David EM, Qiu S, North AJ, Couto CG, Post GS, Waters DJ, Cordon-Cardo C, Hall RD, Gordon BR, Diehl CH, Stenzel KH, Rubin AL. Hydrophilic agarose macrobead cultures select for outgrowth of carcinoma cell populations that can restrict tumor growth. Cancer Res. 2011 Feb 1;71(3):725-35. doi: 10.1158/0008-5472.CAN-10-2258. Epub 2011 Jan 24. PMID 21266362
- [Background] Smith BH, Gazda LS, Conn BL, Jain K, Asina S, Levine DM, Parker TS, Laramore MA, Martis PC, Vinerean HV, David EM, Qiu S, Cordon-Cardo C, Hall RD, Gordon BR, Diehl CH, Stenzel KH, Rubin AL. Three-dimensional culture of mouse renal carcinoma cells in agarose macrobeads selects for a subpopulation of cells with cancer stem cell or cancer progenitor properties. Cancer Res. 2011 Feb 1;71(3):716-24. doi: 10.1158/0008-5472.CAN-10-2254. Epub 2011 Jan 24. PMID 21266363
- [Background] Gazda LS, Martis PC, Laramore MA, Bautista MA, Dudley A, Vinerean HV, Smith BH. Treatment of agarose-agarose RENCA macrobeads with docetaxel selects for OCT4(+) cells with tumor-initiating capability. Cancer Biol Ther. 2013 Dec;14(12):1147-57. doi: 10.4161/cbt.26455. Epub 2013 Sep 12. PMID 24025409
- [Background] Smith BH, Parikh T, Andrada ZP, Fahey TJ, Berman N, Wiles M, Nazarian A, Thomas J, Arreglado A, Akahoho E, Wolf DJ, Levine DM, Parker TS, Gazda LS, Ocean AJ. First-in-Human Phase 1 Trial of Agarose Beads Containing Murine RENCA Cells in Advanced Solid Tumors. Cancer Growth Metastasis. 2016 Aug 2;9:9-20. doi: 10.4137/CGM.S39442. eCollection 2016. PMID 27499645
- [Background] Smith BH, Gazda LS, Fahey TJ, Nazarian A, Laramore MA, Martis P, Andrada ZP, Thomas J, Parikh T, Sureshbabu S, Berman N, Ocean AJ, Hall RD, Wolf DJ. Clinical laboratory and imaging evidence for effectiveness of agarose-agarose macrobeads containing stem-like cells derived from a mouse renal adenocarcinoma cell population (RMBs) in treatment-resistant, advanced metastatic colorectal cancer: Evaluation of a biological-systems approach to cancer therapy (U.S. FDA IND-BB 10091; NCT 02046174, NCT 01053013). Chin J Cancer Res. 2018 Feb;30(1):72-83. doi: 10.21147/j.issn.1000-9604.2018.01.08. PMID 29545721

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited based on physician referral at five academic medical centers between March 2013 and November 2017. The first participant was implanted on April 11, 2014 and the last implant was March 7, 2018.
Pre-assignment Details: 70 participants provided informed consent to participate in the study (Group A n=67; Group B n=3). Of these, 41 mCRC patients were enrolled in the RENCA macrobead implantation arm (Group A) and 3 subjects were enrolled in the Best Supportive Care arm (Group B). The 25 subjects who were not enrolled into Group A, after providing informed consent, had failed the respective eligibility criteria.
Groups:
- Macrobead Implantation Arm: mCRC patients who will undergo up to 4 implantations of RENCA macrobeads (no less than 3 months apart), at a dosage level of 8 RENCA macrobeads per kilogram of body weight.
  RENCA macrobeads
- Best Supportive Care Arm: mCRC patients who had previously decided (independently of this study) to receive, or continue receiving, best supportive care, defined as management of symptoms aimed at maintaining or improving quality of life, but not including approved therapies targeting the patient's malignancy.
Period: Overall Study
Arm/Group | Macrobead Implantation Arm | Best Supportive Care Arm
Started | 42 | 3
Completed | 41 | 3
Not Completed | 1 | 0
Not completed — Too many adhesions to receive implant (at time of surgery). | 1 | 0

BASELINE CHARACTERISTICS:
Population: The analysis population was limited to those in Group A, Macrobead Implantation Arm. Group B, Best Supportive Care, was only able to enroll 3 of 80 participants planned. Per Group B investigators, the entry criteria were flagged as being impossible for reliable enrollment. Therefore, the reported study results are only from participants who were enrolled and implanted with RENCA macrobeads.
Groups:
- Macrobead Implantation Arm: mCRC patients who will undergo up to 4 implantations of RENCA macrobeads (no less than 3 months apart), at a dosage level of 8 RENCA macrobeads per kilogram of body weight.
Arm/Group | Macrobead Implantation Arm
Number analyzed (Participants) | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.9 (14.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 20
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 33
  African American | 4
  Hispanic | 3
  Asian | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 41

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: The primary objective of this study was to evaluate the efficacy of RENCA macrobead implantation as assessed by overall survival in subjects with treatment-resistant mCRC.
Time Frame: From date of the most recent scan prior to the first macrobead implantation; assessed up to 32 months.
Population: The analysis population was limited to those in Group A, Macrobead Implantation Arm. Group B, Best Supportive Care, was only able to enroll 3 of 80 participants planned. Per Group B investigators, the entry criteria were flagged as being impossible for reliable enrollment. Therefore, these results focus on the participants who were enrolled and implanted with RENCA macrobeads.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Macrobead Implantation Arm
Number analyzed (Participants) | 41
months | 9.25 [6.03 to 11.44]

2. Secondary Outcome: Performance Status (ECOG Score)
Description: The Eastern Cooperative Oncology Group (ECOG) performance scale is a 5-point scale, where 0 denotes perfect health and 5 is death. It is used by clinicians to assess disease progression and how the disease is affecting the daily living abilities of the patient. The ECOG Performance Status scores are defined as follows:
  * 0: Fully active, able to carry on all pre-disease activities without restriction.
  * 1: Restricted in physical strenuous activity, but ambulatory and able to carry out work of a light or sedentary nature (e.g. light house work, office work).
  * 2: Ambulatory and capable of all self-care, but unable to carry out any work activities, up and about more than 50% of waking hours.
  * 3: Capable of only limited self-care, confined to bed or chair 50% or more of waking hours.
  * 4: Completely disabled, cannot carry on any self-care, totally confined to bed or chair.
  * 5: Death
Time Frame: Baseline; Day 14, 30, 60 post-Implant 1; Day 14, 30, 60 post-Implant 2
Population: Analysis population was limited to the arm "macrobead implantation" as the proposed second arm "best supportive care" did not enroll enough participants to facilitate reliable analysis.
  Implant 1 (day 0 to day 60): Participants who received at least one RENCA macrobead implantation; Implant 2 (day 0 to day 60): Participants who received at least two RENCA macrobead implantations.
Measure: Count of Participants; unit: Participants
Groups:
- Implant 1: Day 0: ECOG score at day 0 of first implantation
- Implant 1: Day 14: ECOG score at day 14 after first implantation
- Implant 1: Day 30: ECOG score at day 30 following first implantation
- Implant 1: Day 60: ECOG score at day 60 following first implantation
- Implant 2: Day 0: ECOG score at day 0 of second implantation
- Implant 2: Day 14: ECOG score at day 14 following second implantation
- Implant 2: Day 30: ECOG score at day 30 following second implantation
- Implant 2: Day 60: ECOG score at day 60 following second implantation
Arm/Group | Implant 1: Day 0 | Implant 1: Day 14 | Implant 1: Day 30 | Implant 1: Day 60 | Implant 2: Day 0 | Implant 2: Day 14 | Implant 2: Day 30 | Implant 2: Day 60
Number analyzed (Participants) | 41 | 38 | 36 | 27 | 8 | 8 | 7 | 7
Participants
  ECOG Score 0 | 16 | 5 | 5 | 11 | 5 | 4 | 4 | 4
  ECOG Score 1 | 21 | 23 | 23 | 8 | 2 | 3 | 2 | 2
  ECOG Score 2 | 4 | 7 | 7 | 7 | 1 | 1 | 1 | 1
  ECOG Score 3 | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 0
  ECOG Score 4 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  ECOG Score 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: Activities of Daily Living (KPS Score)
Description: Karnofsky Performance Status (KPS) is a self-rated scale that measures the participant's ability to perform daily functions, ranging from 0 ("dead") to 100 ("normal, no complaints, no evidence of disease). Karnofsky scores are defined as follows:
  * 100: Normal; no complaints; no evidence of disease
  * 90: Able to carry on normal activity with effort, minor sign or symptoms of disease
  * 80: Normal activity with effort; some sign or symptoms of disease
  * 70: Cares for self; unable to carry on normal activity or do active work
  * 60: Requires occasional assistance, but is able to care for most personal needs
  * 50: Requires considerable assistance and frequent medical care
  * 40: Disabled; requires special care and assistance
  * 30: Severely disabled; hospitalization is indicated, although death is not imminent
  * 20: Very sick; hospitalization/active support treatment is necessary
  * 10: Moribund; fatal processes progressively worsening
  * 0: Dead
Time Frame: Baseline; Day 14, 30, 60 post-Implant 1; Day 14, 30, 60 post-Implant 2
Population: Analysis population was limited to the arm "macrobead implantation" as the proposed second arm "best supportive care" did not enroll enough participants to facilitate reliable analysis. Implant 1 (Day 0 to Day 60): Participants who had received at least 1 RENCA macrobead implantation; Implant 2 (Day 0 to Day 60): Participants who had received at least 2 RENCA macrobead implantations.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Implant 1: Day 0: KPS score at pre-screening for first implantation
- Implant 1: Day 14: KPS score at day 14 after first implantation
- Implant 1: Day 30: KPS score at day 30 following first implantation
- Implant 1: Day 60: KPS score at day 60 following first implantation
- Implant 2: Day 0: KPS score at pre-screening for second implantation (day 90 following first implantation).
- Implant 2: Day 14: KPS score at day 14 following second implantation
- Implant 2: Day 30: KPS score at day 30 following second implantation
- Implant 2: Day 60: KPS score at day 60 following second implantation
Arm/Group | Implant 1: Day 0 | Implant 1: Day 14 | Implant 1: Day 30 | Implant 1: Day 60 | Implant 2: Day 0 | Implant 2: Day 14 | Implant 2: Day 30 | Implant 2: Day 60
Number analyzed (Participants) | 40 | 39 | 34 | 26 | 7 | 8 | 7 | 7
score on a scale | 88.3 (9.6) | 82.1 (13.6) | 74.3 (23.7) | 81.8 (19.1) | 94.3 (5.4) | 83.3 (16.7) | 93.3 (7.7) | 91.4 (9.9)

4. Secondary Outcome: Global Health Status
Description: The European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ-C30, version 3.0) consists of 30 questions which pertain to: five functional scales, three symptom scales, a global health status score, and six single items.
  The Global Health Status is assessed from 2 of the 30 questions (Question 29 and 30), whose response score ranges on a 7 point scale. The score for physical function is calculated based on the average score from these 2 questions. A linear transformation is used to standardize these responses. Using this linear transformation, the minimum value is 0 (worst outcome, poor) and the maximum value is 100 (best outcome, excellent). Therefore, increasing values indicate better outcome and decreasing values indicate worse outcome.
Time Frame: Baseline; Day 14, 30, 60 post-Implant 1; Day 14, 30, 60 post-Implant 2
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Implant 1: Day 0: Global health score at pre-screening for first implantation
- Implant 1: Day 14: Global health score at day 14 after first implantation
- Implant 1: Day 30: Global health score at day 30 following first implantation
- Implant 1: Day 60: Global health score at day 60 following first implantation
- Implant 2: Day 0: Global health score at pre-screening for second implantation (day 90 following first implantation)
- Implant 2: Day 14: Global health score at day 14 following second implantation
- Implant 2: Day 30: Global health score at day 30 following second implantation
- Implant 2: Day 60: Global health score at day 60 following second implantation
Arm/Group | Implant 1: Day 0 | Implant 1: Day 14 | Implant 1: Day 30 | Implant 1: Day 60 | Implant 2: Day 0 | Implant 2: Day 14 | Implant 2: Day 30 | Implant 2: Day 60
Number analyzed (Participants) | 41 | 39 | 34 | 26 | 8 | 8 | 7 | 7
score on a scale | 68.70 (22.03) | 50.21 (24.37) | 56.13 (29.61) | 69.87 (28.48) | 84.38 (17.50) | 75.00 (14.77) | 83.33 (11.79) | 83.33 (26.79)

5. Secondary Outcome: Physical Function
Description: TThe European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ-C30, version 3.0) consists of 30 questions which pertain to: five functional scales (including physical function), three symptom scales, a global health status score, and six single items.
  Physical Function is assessed from 5 of the 30 questions (Questions 1-5), whose response score ranges on a 4 point scale. The score for physical function is calculated based on the average score from these 5 questions. A linear transformation is used to standardize these responses. Using this linear transformation, the minimum value is 0 (worst outcome, poor functionality) and the maximum value is 100 (best outcome, better functionality). Therefore, increasing values indicate better outcome and decreasing values indicate worse outcome.
Time Frame: Baseline; Day 14, 30, 60 post-Implant 1; Day 14, 30, 60 post-Implant 2
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Implant 1: Day 0: EORTC/Physical functioning score at pre-screening for first implantation
- Implant 1: Day 14: EORTC/Physical functioning score at day 14 following first implantation
- Implant 1: Day 30: EORTC/Physical functioning score at day 30 following first implantation
- Implant 1: Day 60: EORTC/Physical functioning score at day 60 following first implantation
- Implant 2: Day 0: EORTC/Physical functioning score at pre-screening for second implantation (day 90 following first implantation).
- Implant 2: Day 14: EORTC/Physical functioning score at day 14 following second implantation
- Implant 2: Day 30: EORTC/Physical functioning score at day 30 following second implantation
- Implant 2: Day 60: EORTC/Physical functioning score at day 60 following second implantation
Arm/Group | Implant 1: Day 0 | Implant 1: Day 14 | Implant 1: Day 30 | Implant 1: Day 60 | Implant 2: Day 0 | Implant 2: Day 14 | Implant 2: Day 30 | Implant 2: Day 60
Number analyzed (Participants) | 41 | 39 | 36 | 26 | 8 | 8 | 7 | 6
score on a scale | 80.65 (17.94) | 69.57 (24.79) | 82.50 (12.96) | 83.50 (14.13) | 91.67 (9.26) | 90.00 (9.26) | 92.90 (4.88) | 90.00 (6.32)

6. Secondary Outcome: Role Function
Description: The European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ-C30, version 3.0) consists of 30 questions which pertain to: five functional scales (including role function), three symptom scales, a global health status score, and six single items.
  Role Function is assessed from 2 of the 30 questions (Questions 6 and 7), whose response score ranges on a 4 point scale. The score for role function is calculated based on the average score from these 2 questions. A linear transformation is used to standardize these responses. Using this linear transformation, the minimum value is 0 (worst outcome, poor functionality) and the maximum value is 100 (best outcome, better functionality). Therefore, increasing values indicate better outcome and decreasing values indicate worse outcome.
Time Frame: Baseline; Day 14, 30, 60 post-Implant 1; Day 14, 30, 60 post-Implant 2
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Implant 1: Day 0: EORTC/Role functioning score at pre-screening for first implantation
- Implant 1: Day 14: EORTC/Role functioning score at day 14 following first implantation
- Implant 1: Day 30: EORTC/Role functioning score at day 30 following first implantation
- Implant 1: Day 60: EORTC/Role functioning score at day 60 following first implantation
- Implant 2: Day 0: EORTC/Role functioning score at pre-screening for second implantation (day 90 following first implantation).
- Implant 2: Day 14: EORTC/Role functioning score at day 14 following second implantation
- Implant 2: Day 30: EORTC/Role functioning score at day 30 following second implantation
- Implant 2: Day 60: EORTC/Role functioning score at day 60 following second implantation
Arm/Group | Implant 1: Day 0 | Implant 1: Day 14 | Implant 1: Day 30 | Implant 1: Day 60 | Implant 2: Day 0 | Implant 2: Day 14 | Implant 2: Day 30 | Implant 2: Day 60
Number analyzed (Participants) | 41 | 39 | 34 | 26 | 8 | 8 | 7 | 7
score on a scale | 81.71 (20.00) | 55.56 (32.07) | 61.27 (32.75) | 74.36 (30.99) | 89.58 (15.27) | 60.42 (43.59) | 85.71 (20.25) | 95.24 (12.59)

7. Secondary Outcome: Emotional Function
Description: The European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ-C30, version 3.0) consists of 30 questions which pertain to: five functional scales (including emotional function), three symptom scales, a global health status score, and six single items.
  Emotional Function is assessed from 4 of the 30 questions (Questions 21-24), whose response score ranges on a 4 point scale. The score for role function is calculated based on the average score from these 4 questions. A linear transformation is used to standardize these responses. Using this linear transformation, the minimum value is 0 (worst outcome, poor functionality) and the maximum value is 100 (best outcome, better functionality). Therefore, increasing values indicate better outcome and decreasing values indicate worse outcome.
Time Frame: Baseline; Day 14, 30, 60 post-Implant 1; Day 14, 30, 60 post-Implant 2
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Implant 1: Day 0: EORTC/Emotional functioning score at pre-screening for first implantation
- Implant 1: Day 14: EORTC/Emotional functioning score at day 14 following first implantation
- Implant 1: Day 30: EORTC/Emotional functioning score at day 30 following first implantation
- Implant 1: Day 60: EORTC/Emotional functioning score at day 60 following first implantation
- Implant 2: Day 0: EORTC/Emotional functioning score at pre-screening for second implantation (day 90 following first implantation).
- Implant 2: Day 14: EORTC/Emotional functioning score at day 14 following second implantation
- Implant 2: Day 30: EORTC/Emotional functioning score at day 30 following second implantation
- Implant 2: Day 60: EORTC/Emotional functioning score at day 60 following second implantation
Arm/Group | Implant 1: Day 0 | Implant 1: Day 14 | Implant 1: Day 30 | Implant 1: Day 60 | Implant 2: Day 0 | Implant 2: Day 14 | Implant 2: Day 30 | Implant 2: Day 60
Number analyzed (Participants) | 41 | 39 | 34 | 26 | 8 | 8 | 7 | 7
score on a scale | 79.07 (22.06) | 72.65 (28.74) | 76.23 (27.91) | 80.56 (20.79) | 86.46 (11.73) | 78.13 (19.89) | 83.33 (19.84) | 88.10 (15.11)

8. Secondary Outcome: Cognitive Function
Description: The European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ-C30, version 3.0) consists of 30 questions which pertain to: five functional scales (including cognitive function), three symptom scales, a global health status score, and six single items.
  Cognitive Function is assessed from 2 of the 30 questions (Question 20 and 25), whose response score ranges on a 4 point scale. The score for role function is calculated based on the average score from these 2 questions. A linear transformation is used to standardize these responses. Using this linear transformation, the minimum value is 0 (worst outcome, poor functionality) and the maximum value is 100 (best outcome, better functionality). Therefore, increasing values indicate better outcome and decreasing values indicate worse outcome.
Time Frame: Baseline; Day 14, 30, 60 post-Implant 1; Day 14, 30, 60 post-Implant 2
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Implant 1: Day 0: EORTC/Cognitive functioning score at pre-screening for first implantation
- Implant 1: Day 14: EORTC/Cognitive functioning score at day 14 following first implantation
- Implant 1: Day 30: EORTC/Cognitive functioning score at day 30 following first implantation
- Implant 1: Day 60: EORTC/Cognitive functioning score at day 60 following first implantation
- Implant 2: Day 0: EORTC/Cognitive functioning score at pre-screening for second implantation (day 90 following first implantation).
- Implant 2: Day 14: EORTC/Cognitive functioning score at day 14 following second implantation
- Implant 2: Day 30: EORTC/Cognitive functioning score at day 30 following second implantation
- Implant 2: Day 60: EORTC/Cognitive functioning score at day 60 following second implantation
Arm/Group | Implant 1: Day 0 | Implant 1: Day 14 | Implant 1: Day 30 | Implant 1: Day 60 | Implant 2: Day 0 | Implant 2: Day 14 | Implant 2: Day 30 | Implant 2: Day 60
Number analyzed (Participants) | 41 | 39 | 34 | 26 | 8 | 8 | 7 | 7
score on a scale | 83.74 (16.02) | 83.76 (21.46) | 85.78 (15.43) | 86.54 (16.34) | 93.75 (12.40) | 90.15 (13.27) | 97.62 (6.29) | 95.24 (8.13)

9. Secondary Outcome: Social Function
Description: The European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ-C30, version 3.0) consists of 30 questions which pertain to: five functional scales (including social function), three symptom scales, a global health status score, and six single items.
  Social Function is assessed from 2 of the 30 questions (Question 26 and 27), whose response score ranges on a 4 point scale. The score for role function is calculated based on the average score from these 2 questions. A linear transformation is used to standardize these responses. Using this linear transformation, the minimum value is 0 (worst outcome, poor functionality) and the maximum value is 100 (best outcome, better functionality). Therefore, increasing values indicate better outcome and decreasing values indicate worse outcome.
Time Frame: Baseline; Day 14, 30, 60 post-Implant 1; Day 14, 30, 60 post-Implant 2
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Implant 1: Day 0: EORTC/Social functioning score at pre-screening for first implantation
- Implant 1: Day 14: EORTC/Social functioning score at day 14 following first implantation
- Implant 1: Day 30: EORTC/Social functioning score at day 30 following first implantation
- Implant 1: Day 60: EORTC/Social functioning score at day 60 following first implantation
- Implant 2: Day 0: EORTC/Social functioning score at pre-screening for second implantation (day 90 following first implantation).
- Implant 2: Day 14: EORTC/Social functioning score at day 14 following second implantation
- Implant 2: Day 30: EORTC/Social functioning score at day 30 following second implantation
- Implant 2: Day 60: EORTC/Social functioning score at day 60 following second implantation
Arm/Group | Implant 1: Day 0 | Implant 1: Day 14 | Implant 1: Day 30 | Implant 1: Day 60 | Implant 2: Day 0 | Implant 2: Day 14 | Implant 2: Day 30 | Implant 2: Day 60
Number analyzed (Participants) | 41 | 39 | 34 | 26 | 8 | 8 | 7 | 7
score on a scale | 76.83 (22.63) | 67.52 (33.21) | 69.61 (26.74) | 78.85 (26.89) | 93.75 (8.63) | 93.75 (12.40) | 88.10 (20.89) | 90.48 (13.11)

10. Secondary Outcome: Pain Assessment
Description: Participants were asked to rate their pain on a discrete scale (from 0 = "no pain" to 100 "worst pain imaginable, unbearable"). The worst pain at each time point was used in the analysis.
Time Frame: Baseline; Day 14, 30, 60 post-Implant 1; Day 14, 30, 60 post-Implant 2
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Implant 1: Day 0: Pain Assessment score at pre-screening for first implantation
- Implant 1: Day 14: Pain Assessment score at day 14 following first implantation
- Implant 1: Day 30: Pain Assessment score at day 30 following first implantation
- Implant 1: Day 60: Pain Assessment score at day 60 following first implantation
- Implant 2: Day 0: Pain Assessment score at pre-screening for second implantation (day 90 following first implantation).
- Implant 2: Day 14: Pain Assessment score at day 14 following second implantation
- Implant 2: Day 30: Pain Assessment score at day 30 following second implantation
- Implant 2: Day 60: Pain Assessment score at day 60 following second implantation
Arm/Group | Implant 1: Day 0 | Implant 1: Day 14 | Implant 1: Day 30 | Implant 1: Day 60 | Implant 2: Day 0 | Implant 2: Day 14 | Implant 2: Day 30 | Implant 2: Day 60
Number analyzed (Participants) | 41 | 39 | 34 | 26 | 8 | 8 | 7 | 7
score on a scale | 26.83 (26.58) | 52.56 (30.24) | 41.18 (30.22) | 33.33 (33.67) | 16.67 (19.92) | 22.92 (19.79) | 14.29 (20.25) | 14.29 (24.39)

11. Other Pre Specified Outcome: Tumor Marker Response (CEA and CA 19-9)
Description: Tumor markers included serum carcinoembryonic antigen (CEA) and cancer antigen 19-9 (CA 19-9), and were assessed on all participants in the RENCA macrobead implantation arm at baseline and at subsequent evaluation points to further assess tumor response to RENCA macrobead implantation. A tumor marker response was defined as a greater than or equal to 20% decrease in one or both of CEA or CA 19-9.
Time Frame: Change from baseline up to and including day 90 post-Implant 1.
Population: Participants receiving at least one RENCA macrobead implantation whose tumor marker response was greater than or equal to 20% decrease in one or both of CEA or CA 19-9.
Measure: Count of Participants; unit: Participants
Groups:
- CEA Only: Participants whose tumor marker response was greater than or equal to 20% decrease from baseline in CEA only [up to and including day 90 after the first implant).
- CA 19-9 Only: Participants whose tumor marker response was greater than or equal to 20% decrease from baseline in CA 19-9 only [up to and including day 90 after the first implant).
- Both CEA and CA 19-9: Participants whose tumor marker response was greater than or equal to 20% decrease from baseline in both CEA and CA 19-9 [up to and including day 90 after the first implant).
- Non-responder: Participants whose tumor marker response (serum level of CEA and/or CA 19-9) did not decrease by greater than or equal to 20% of baseline value.
Arm/Group | CEA Only | CA 19-9 Only | Both CEA and CA 19-9 | Non-responder
Number analyzed (Participants) | 41 | 41 | 41 | 41
Participants | 6 | 5 | 12 | 18

12. Other Pre Specified Outcome: Overall Survival by Tumor Marker Response
Description: Overall survival (OS) of participants by tumor marker response. A responder is a participant having a decrease from baseline of 20% or more in CEA or CA 19-9 within 90 days of Implant. OS is the time interval between the date of radiographically documented disease progression and the date of death due to any cause. Participants still alive at the end of the study are censored at 22OCT2018.
Time Frame: 30 months
Population: All participants who had received at least one implantation of RENCA macrobeads.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Responder: Responders is defined as any participant having a 20% or more decrease from baseline levels of the biomarker carcinoembryonic antigen (CEA) or cancer antigen 19-9 (CA 19-9), or both, following RENCA macrobead implantation.
- Non-Responder: Non-Responder is defined as any participant not having a 20% or more decrease from baseline levels of the biomarker carcinoembryonic antigen (CEA) or cancer antigen 19-9 (CA 19-9), or both, following RENCA macrobead implantation.
Arm/Group | Responder | Non-Responder
Number analyzed (Participants) | 23 | 18
months | 10.33 [7.05 to 11.51] | 6.82 [3.54 to 14.98]

13. Other Pre Specified Outcome: Necrosis Comparison of Tumors Using PET-CT Scan
Description: Tumors were assessed by positron emission tomography (PET)-CT scan at baseline and day 90 following the first RENCA macrobead implantation. The use of [13]F-fluorodeoxyglucose (FDG) uptake for the detection of lesions >1 cm in diameter allowed evaluation of metabolic activity. Decreases in FDG uptake were indicative of metabolic suppression of the tumor. The use of PET-CT scanning indicated anatomical localization, approximate size/volume of primary tumor and metastatic lesion(s), and assessment of metabolic activity of the tumor (as an indicator of metabolic health and necrosis).
  Disease state is reported as a function of Tumor measurement divided by SUVmax. Changes were assessed between day 90 post RENCA macrobead implant and baseline values. Patients with no change = stable; patients with decreased values = decreased/necrosis, and patients with increased values = increased.
Time Frame: Day 90 post-Implant 1
Population: Participants who had received at least one macrobead implant and for whom baseline PET-CT scan and day 90 post-Implant 1 PET-CT scan data were available.
  n= 26 subjects; 77 lesions evaluated
Measure: Count of Units; unit: lesions
Units Other Than Participants: lesions
Groups:
- Stable Disease: Stable disease based on imaging results [Tumor measurement/SUV max].
- Decreased/Necrosis: Decreased/Necrosis observed based on imaging results [tumor measurement/SUV max].
- Increased: Increased SUVmax, tumor measurement based on imaging results.
Arm/Group | Stable Disease | Decreased/Necrosis | Increased
Number analyzed (Participants) | 26 | 26 | 26
Number analyzed (lesions) | 77 | 77 | 77
lesions | 19 | 37 | 21

ADVERSE EVENTS:
Time Frame: From date of first macrobead implantation; assessed up to 32 months.
Description: The NCI CTCAE was used to standardize the terminology and grade the severity of reported adverse events. The Principal and Sub-Investigators, and the Attending Physicians, were responsible for monitoring adverse events and the safety of all participants. The Data Safety Monitoring Board, independently and in collaboration with the PIs, monitored and reviewed all safety findings, including study status, all SAEs, AEs > Grade 2, laboratory values of special interest and all subject deaths.
Groups:
- Macrobead Implantation Arm: Analysis population was limited to the arm "macrobead implantation" as the proposed second arm "best supportive care" did not enroll enough participants to facilitate reliable analysis. The arm reported here includes all patients who had at least one implantation of RENCA macrobeads.
Arm/Group | Macrobead Implantation Arm
All-Cause Mortality (participants affected / at risk) | 36/41
Serious Adverse Events (participants affected / at risk) | 27/41
Other Adverse Events (participants affected / at risk) | 41/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Macrobead Implantation Arm (N=41)
Anaemia (Blood and lymphatic system disorders) | 2
Leukocytosis (Blood and lymphatic system disorders) | 1
Tachycardia (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 7
Nausea (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 3
Abdominal distension (Gastrointestinal disorders) | 2
Ascites (Gastrointestinal disorders) | 1
Large intestinal obstruction (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1
Disease progression (General disorders) | 7 — General disorders and administration site conditions
Pyrexia (General disorders) | 3 — General disorders and administration site conditions
Fatigue (General disorders) | 1 — General disorders and administration site conditions
Malaise (General disorders) | 1 — General disorders and administration site conditions
Pain (General disorders) | 1 — General disorders and administration site conditions
Peritonitis (Infections and infestations) | 2
Abdominal abscess (Infections and infestations) | 1
Abdominal infection (Infections and infestations) | 1
Empyema (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Spinal column injury (Injury, poisoning and procedural complications) | 1
Activated partial thromboplastin time prolonged (Investigations) | 1
Blood biliriubin increased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Failure to thrive (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Cerebellar tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Depressed level of consciousness (Nervous system disorders) | 1
Dysarthria (Nervous system disorders) | 1
Mental status changes (Psychiatric disorders) | 1
Renal failure acute (Renal and urinary disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Macrobead Implantation Arm (N=41)
Anaemia (Blood and lymphatic system disorders) | 5
Abdominal pain (Gastrointestinal disorders) | 15
Nausea (Gastrointestinal disorders) | 15
Constipation (Gastrointestinal disorders) | 14
Diarrhoea (Gastrointestinal disorders) | 14
Abdominal distension (Gastrointestinal disorders) | 11
Vomiting (Gastrointestinal disorders) | 10
Flatulence (Gastrointestinal disorders) | 4
Abdominal pain, upper (Gastrointestinal disorders) | 3
Ascites (Gastrointestinal disorders) | 2
Proctalgia (Gastrointestinal disorders) | 3
Fatigue (General disorders) | 19 — General disorders and administration site conditions
Pyrexia (General disorders) | 9 — General disorders and administration site conditions
Oedema peripheral (General disorders) | 7 — General disorders and administration site conditions
Asthenia (General disorders) | 5 — General disorders and administration site conditions
Chills (General disorders) | 3 — General disorders and administration site conditions
Gait disturbance (General disorders) | 3 — General disorders and administration site conditions
Urinary tract infection (Infections and infestations) | 3
Incision site pain (Injury, poisoning and procedural complications) | 9
Weight decreased (Investigations) | 6
Activated partial thromboplastin time prolonged (Investigations) | 4
International normalised ratio increased (Investigations) | 3
Decreased appetite (Metabolism and nutrition disorders) | 17
Dehydration (Metabolism and nutrition disorders) | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 5
Hypoalbuminaemia (Metabolism and nutrition disorders) | 5
Abdominal discomfort (Gastrointestinal disorders) | 2
Abdominal pain, lower (Gastrointestinal disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 2
Contusion (Injury, poisoning and procedural complications) | 2
Fall (Injury, poisoning and procedural complications) | 2
Incision site complication (Injury, poisoning and procedural complications) | 2
Blood alkaline phosphatase, increased (Investigations) | 2
Blood creatinine, increased (Investigations) | 2
Hypokalaemia (Metabolism and nutrition disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 7
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 5
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Flank Pain (Musculoskeletal and connective tissue disorders) | 2
Headache (Nervous system disorders) | 5
Dizziness (Nervous system disorders) | 4
Lethargy (Nervous system disorders) | 3
Disturbance in attention (Nervous system disorders) | 2
Insomnia (Psychiatric disorders) | 4
Agitation (Psychiatric disorders) | 3
Confusional state (Psychiatric disorders) | 3
Anxiety (Psychiatric disorders) | 2
Restlessness (Psychiatric disorders) | 2
Dysuria (Renal and urinary disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 5
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 5
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2
Night sweats (Skin and subcutaneous tissue disorders) | 4
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3
Uticaria (Skin and subcutaneous tissue disorders) | 2
Deep vein thrombosis (Vascular disorders) | 2

LIMITATIONS AND CAVEATS:
Group B was only able to enroll 3/80 participants planned for the best supportive care management arm of this study. As per Group B investigators, the entry criteria were flagged as being impossible for reliable enrollment. Therefore, the results reported here focus on the Group A participants, those which were implanted with RENCA macrobeads.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor retains the first right for scientific disclosure of study results. PI may draft a study results disclosure for scientific publication following the earlier of sponsor's disclosure or 12 months after study completion at all sites. Sponsor has 60 days to review PI's draft for patentable subject matter or confidential information. PI will delete any confidential information and delay any disclosure for another 60 days for sponsor to secure proprietary protection.

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-01-25): https://cdn.clinicaltrials.gov/large-docs/74/NCT02046174/SAP_000.pdf
  • Study Protocol (2013-12-23): https://cdn.clinicaltrials.gov/large-docs/74/NCT02046174/Prot_001.pdf